CLINICAL TRIAL: NCT01152060
Title: an Open Parallel Clinical Trial in HBV-GN Patients
Brief Title: Treatment for HBV-MN Patients in Chinese: An Open Parallel Controlled Trial
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nanchang University (Other)
Responsible Party: ethics committee of Nanchang University, second affiliated hospital
Other Study IDs: NCT00100504
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-05

CONDITIONS: Proteinuria; HBVe-antigen
Keywords: remission of proteinuria; HBVe-antigen
MeSH Terms: conditions — Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- prednisone
- prednisone and anti-virus

SUMMARY:
Lamivudine treatment for HBV-DNA negative HBV-GN patients.

DETAILED DESCRIPTION:
lamivudine and predinisone treatment for HBV-DNA negative HBV-GN patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult HBV-GN patients with biopsy-proven MN, heavy protinuria, HBsAg or HBeAg positive, HBV-DNA negative

Exclusion Criteria:

* Primary MN patients, HBV-DNA positive

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HBV-MN patients with heavy proteinuria in adults; HBsAg or HBeAg positive; HBV-DNA negative
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gaosi XU, MD & PhD, Study Director — second affiliated hospital to nanchang university

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952
- [Derived] Xu G, Duang Z, Wu X, Zou H, Fang X, Tu W. Treatment of hepatitis B virus-associated membranous nephritis patients in Chinese: an open parallel controlled trial. Clin Chem Lab Med. 2011 Jun;49(6):1077-8. doi: 10.1515/CCLM.2011.168. Epub 2011 Mar 17. No abstract available. PMID 21410411